CLINICAL TRIAL: NCT04177056
Title: Stereotactic Body Radiotherapy for Osseous Low Alpha-Beta Resistant Metastases for Pain Relief
Acronym: SOLAR-P
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hamilton Health Sciences Corporation (Other)
Collaborators: Juravinski Cancer Centre Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 7905
Record Dates: First submitted 2019-11-14; First posted 2019-11-26 (Actual); Last update posted 2021-08-02 (Actual); Status verified 2021-07

CONDITIONS: Bone Metastases; Prostate Cancer; Breast Cancer; Renal Cell Carcinoma; Melanoma
Keywords: SOLAR-P; SBRT; Bone metastases; stereotactic; pain relief; quality of life; palliation; low alpha beta; radioresistant
MeSH Terms: conditions — Prostatic Neoplasms; Breast Neoplasms; Carcinoma, Renal Cell; Melanoma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Stereotactic Body Radiotherapy (Experimental): High dose SBRT to lesion(s) of interest.
  Interventions: Radiation: SBRT

INTERVENTIONS:
Radiation: SBRT — Patients will received a single fraction of 15-20 Gy to bone metastases causing pain. Planning and delivery will be conducted using a volumetric modulated arc therapy (VMAT) approach on the Varian TrueBeam platform. Patients will be CT simulated, with vac-lock immobilization. Use of 4-dimensional CT will be dependent on the area being treated. Daily image guidance will be performed using cone beam CT aligning to relevant bony anatomy.

SUMMARY:
Radiation therapy has been shown to be very effective at relieving pain caused by bone metastases. However, certain types of cancers such as prostate, breast, kidney, and melanoma can have resistance to radiation, making treatment less successful. Stereotactic body radiotherapy (SBRT) is a newer form of focused treatment that gives higher doses of radiation without damage to surrounding organs. It often is used to help control and cure disease, but less commonly as a way to palliate and treat symptoms. This study is looking at using SBRT for the purposes of improving pain caused by bone metastases in prostate cancer, breast cancer, kidney cancer, and melanoma patients. It is theorized that the higher levels of radiation may be able to combat the resistance some tumour cells have to radiotherapy and provide improved pain response to treatment. The investigators are looking to show that SBRT has a role in helping this group of patients deal with painful bone lesions from their cancer without increasing side effects and toxicity from the radiation treatment.

DETAILED DESCRIPTION:
Stereotactic body radiotherapy (SBRT) has shown promising early results in the management of bone metastases. However, there is a paucity of prospective data studying the use of SBRT for bone metastases originating from low alpha-beta tumors, with systematic reporting of changes in pain scores and analgesia use over time. The vast majority data looking at SBRT in bone lesions focuses on local control and survival, rather than more tangible outcomes in a palliative population including symptomatic control, durability of response, and patient reported quality of life; a component that is understudied in this group despite its tremendous value. Furthermore, SBRT for bone metastases has yet to become common practice given the limited evidence for its efficacy and uncertainty in regards to toxicity.

The current study proposes an investigation of the potential benefits of SBRT for symptomatic bone metastases in patients with prostate cancer, breast cancer, renal cell carcinoma, melanoma, and sarcoma. The investigators look to conduct a prospective cohort study that is adequately powered to analyse efficacy in alleviating pain from bone lesions and compare this to well-established rates in literature for conventionally fractionated palliative RT. Furthermore, this study will assess the tolerability of this modality, toxicity rates, and effect on quality of life. If the results show that SBRT has a significant benefit on this population, the goal would be to pursue a larger randomized trial to confirm the findings.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of prostate cancer, renal cell carcinoma, or melanoma
* Radiographic evidence of bone metastases requiring treatment for pain
* Brief Pain Inventory score of ≥ 2

Exclusion Criteria:

* Spinal lesions
* Severe or progressive neurological deficit
* Impending or existing pathological fracture
* Bone metastasis in a previously irradiated site
* Active systemic therapy
* >5 lesions requiring treatment
* Lesions >5 cm in largest diameter
* Life expectancy < 3 months
* Age < 18
* Karnofsky Performance Status < 50
* Unable to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-12-04 (Actual); Primary Completion 2022-03-01 (Estimated); Study Completion 2023-01-01 (Estimated)

PRIMARY OUTCOMES:
Overall Pain Response | 3 months after treatment
  Assessed using the Brief Pain Inventory

SECONDARY OUTCOMES:
Overall Pain Response | 6 months after treatment
  Assessed using the Brief Pain Inventory
Acute Toxicity | 3 months or less
  According to the Common Terminology Criteria for Adverse Events 5.0
Late Toxicity | greater than 3 months
  According to the Common Terminology Criteria for Adverse Events 5.0
Patient-reported Quality of Life | 1 month, 3 months, and 6 months
  Assessed by EORTC quality of life questionnaires
Local Control | up to 1 year
  Assessed radiographically
Rate of Reirradiation/Salvage Surgery | up to 1 year
  Due to instability or symptomatic progression

CONTACTS AND LOCATIONS:
Overall Officials: Anand Swaminath, MD, Principal Investigator — Hamilton Health Sciences Corporation
Locations (1):
- Juravinski Cancer Centre, Hamilton, Ontario, Canada

REFERENCES:
- [Derived] Nguyen EK, Quan K, Parpia S, Tran S, Swaminath A. Stereotactic body radiotherapy for osseous low alpha-beta resistant metastases for pain relief-SOLAR-P. Radiat Oncol. 2021 Sep 3;16(1):170. doi: 10.1186/s13014-021-01897-0. PMID 34479581

DOCUMENTS (1):
  • Study Protocol (2020-11-24): https://cdn.clinicaltrials.gov/large-docs/56/NCT04177056/Prot_000.pdf